CLINICAL TRIAL: NCT00003895
Title: A Randomized Phase II Trial to Determine the Immune Response to a Mutated gp100 Melanoma Peptide (209-2M) Vaccine in HLA-A2 Positive Patients With a >1mm Melanoma on Initial Biopsy
Brief Title: Vaccine Therapy in Treating HLA-A2 Positive Patients With Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02096; NCI-2013-02096 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000067065; NCI-T98-0081; PPMC-IRB-99-9 (Other: Providence Portland Medical Center); 99-9 (Other: Providence Portland Medical Center); T98-0081 (Other: CTEP); R21CA082614 (NIH); NCT02009657 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-07-18 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2016-12

CONDITIONS: Recurrent Melanoma; Stage IA Melanoma; Stage IB Melanoma; Stage IIA Melanoma; Stage IIB Melanoma; Stage IIC Melanoma; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma
MeSH Terms: conditions — Melanoma

ARMS (2):
- gp100:209-217(210M) + HPV 16 E7:12-20 (every 2 weeks) (Experimental): Patients receive gp100:209-217(210M) peptide vaccine and HPV 16 E7:12-20 peptide vaccine mixed with incomplete Freund's adjuvant SC every 2 weeks for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo laboratory biomarker analysis.
  Interventions: Biological: HPV 16 E7:12-20; Biological: gp100:209-217(210M); Other: laboratory biomarker analysis
- gp100:209-217(210M) + HPV 16 E7:12-20 (every 3 weeks) (Experimental): Patients receive gp100:209-217(210M) peptide vaccine and HPV 16 E7:12-20 peptide vaccine mixed with incomplete Freund's adjuvant SC every 3 weeks for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo laboratory biomarker analysis.
  Interventions: Biological: HPV 16 E7:12-20; Biological: gp100:209-217(210M); Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: HPV 16 E7:12-20 — Given SC
Biological: gp100:209-217(210M) — Given SC
  Other Names: G9 209-2M
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized pilot phase II trial studies how well vaccine therapy works in treating human leukocyte antigen class 1 histocompatibility, A-2 (HLA-A2) positive patients with melanoma. Vaccines made from peptides may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the toxicity of administration of gp100: 209-217 (210M) (gp100:209-217[210M] peptide vaccine) and the human papillomavirus (HPV) 16 E7(12-20) peptide (HPV16E7:12-20 peptide vaccine), with adjuvant Montanide ISA-51 (incomplete Freund's adjuvant), to patients who present with a primary melanoma > 1 mm thick.

II. To measure the T-cell response to the modified self-gp100: 209-217 (210M) peptide and the unmodified parental glycoprotein 100 (gp100) peptide.

III. To measure the T-cell response to the control human leukocyte antigen (HLA)-A2.1 restricted cytotoxic T-lymphocyte (CTL) epitope of papilloma virus HPV16E7:12-20.

IV. To determine whether analysis of antigen-specific T-cells using specific HLA-A2/peptide tetramers is an effective method for monitoring the immune response of patients undergoing peptide vaccination and to compare it to enzyme-linked immunosorbent spot (ELISPOT), limiting dilution analysis (LDA) and measurement of intracellular cytokine production (fastimmune).

V. To determine whether there is a difference between the induction of primary peptide-specific T-cell immune responses to the self gp100 peptide versus the foreign E7 peptide.

VI. To compare the immune response induced by vaccinating every 2 weeks for 6 months (a total of 13 vaccinations) vs. every 3 weeks for 6 months (a total of 9 vaccinations).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive gp100:209-217(210M) peptide vaccine and HPV16E7:12-20 peptide vaccine mixed with incomplete Freund's adjuvant subcutaneously (SC) every 2 weeks for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive gp100:209-217(210M) peptide vaccine and HPV16E7:12-20 peptide vaccine mixed with incomplete Freund's adjuvant SC every 3 weeks for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.

In both arms, patients undergo sentinel lymph node biopsy approximately 10 days after the second vaccination. Patients with positive lymph nodes undergo complete lymph node dissection and resume vaccinations.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed primary melanoma of Breslow thickness 1.0-4.0 mm; patients who have had only their initial biopsy are preferred; however, those who have already undergone a wide local excision are also eligible; patients may be enrolled up to three months after their wide local excision
* Patients whose melanoma is > 4.0 mm thick who have positive or negative regional lymph nodes are also eligible
* After accrual to the original 26 patient goal, all patients must be enrolled prior to sentinel lymph node dissection; patients with previous lymph node dissection will not be eligible
* Patients must be HLA typed and be shown to be HLA-A2.1+ by either serologic techniques, flow cytometry, or molecular techniques
* Patients must be ambulatory with good performance status (Karnofsky performance status [PS] 80-100)
* White blood cell (WBC) >= 3500/mm^3
* Platelets (Plt) >= 100,000/mm^3
* Hemoglobin >= 9 gm/100 ml
* Serum creatinine =< 2 mg/dl
* Total bilirubin =< 2.0 mg/dl
* Patients must have recovered from any effects of major surgery and be free of significant systemic infection
* Patients must be negative for human immunodeficiency virus (HIV) antibody by enzyme-linked immunosorbent assay (ELISA) (or negative by Western blot if ELISA is positive) if they are considered to be at high risk; others do not require serologic testing if there are no symptoms or risk factors for HIV disease
* Women of childbearing potential must have a negative pregnancy test and should avoid becoming pregnant while on treatment
* Patients must give written informed consent prior to initiation of therapy; patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy

Exclusion Criteria:

* Patients must not have clinically detectable distant metastases
* Patients who require or are likely to require systemic corticosteroids for intercurrent illness
* Patients with any significant medical disease other than the malignancy (e.g. chronic obstructive pulmonary disorder [COPD], patients with ascites or pleural effusions) which in the opinion of the investigator would significantly increase the risk of immunotherapy
* Patient should be free of any other cancers or deemed at low risk for their recurrence

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1999-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter J. Urba, MD, PhD, Principal Investigator — Providence Cancer Center, Earle A. Chiles Research Institute, Robert W. Franz Cancer Center
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- gp100:209-217(210M)and HPV 16 E7:12-20 (Every 2 Weeks): Patients receive gp100:209-217(210M) peptide vaccine and HPV 16 E7:12-20 peptide vaccine mixed with incomplete Freund's adjuvant SC every 2 weeks for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.
  HPV 16 E7:12-20 peptide vaccine: Given SC
  gp100:209-217(210M) peptide vaccine: Given SC
  laboratory biomarker analysis: Correlative studies
- gp100:209-217(210M) and HPV 16 E7:12-20 (Every 3 Weeks): Patients receive gp100:209-217(210M) peptide vaccine and HPV 16 E7:12-20 peptide vaccine mixed with incomplete Freund's adjuvant SC every 3 weeks for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.
  HPV 16 E7:12-20 peptide vaccine: Given SC
  gp100:209-217(210M) peptide vaccine: Given SC
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | gp100:209-217(210M)and HPV 16 E7:12-20 (Every 2 Weeks) | gp100:209-217(210M) and HPV 16 E7:12-20 (Every 3 Weeks)
Started | 18 | 18
Completed | 11 | 14
Not Completed | 7 | 4
Not completed — Adverse Event | 4 | 0
Not completed — Lack of Efficacy | 1 | 1
Not completed — Patient Vacation | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Every 2 Weeks) | Arm B (Every 3 Weeks) | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 4 | 4 | 8
Gender [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: T Cell Immunity to gp100 Peptide and to E7 12-20 Papilloma Virus Peptide
Description: Frequency measures obtained from each assay will be transformed to (common) logs for purposes of analysis. Repeated measures analyses will be performed on longitudinal data to assess patients' immune response profiles over time. Comparability of assay methods will be assessed with correlation analyses, regression analyses, standard parametric and nonparametric tests, and agreement methods.
  Pre- and post-immunization T-cell immunity to g209-2M peptide, to HPV16E7 peptide, and to a negative control HLA-A2 HIV peptide (pol) were assessed using HLA-A2/peptide tetramer-specific binding analysis. Within-subject analyses were performed to determine differences between pre- and postimmunization responses to the g209 -2M and HPV peptides and to the negative control HIV peptide after completion of 6 months of vaccination. Pre- versus postimmunization response differences were used as criterion measures in between-group (among subjects) analyses.
Time Frame: Baseline to 6 months
Population: Patients were randomly assigned to two different vaccination schedules: group A received vaccinations every 2 weeks for 6 months (13 total injections), and group B received vaccinations every 3 weeks for 6 months (nine total vaccinations).
Measure: Mean (90% Confidence Interval); unit: % of CD8+ T cells
Groups:
- Arm A (Every 2 Weeks, gp100:209-217(210M) and HPV 16 E7:12-20): Patients receive gp100:209-217(210M) peptide vaccine and HPV 16 E7:12-20 peptide vaccine mixed with incomplete Freund's adjuvant SC every 2 weeks for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.
  HPV 16 E7:12-20 peptide vaccine: Given SC
  gp100:209-217(210M) peptide vaccine: Given SC
  laboratory biomarker analysis: Correlative studies
- Arm B (Every 3 Weeks, gp100:209-217(210M) + HPV 16 E7:12-20): Patients receive gp100:209-217(210M) peptide vaccine and HPV 16 E7:12-20 peptide vaccine mixed with incomplete Freund's adjuvant SC every 3 weeks for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.
  HPV 16 E7:12-20 peptide vaccine: Given SC
  gp100:209-217(210M) peptide vaccine: Given SC
  laboratory biomarker analysis: Correlative studies
Arm/Group | Arm A (Every 2 Weeks, gp100:209-217(210M) and HPV 16 E7:12-20) | Arm B (Every 3 Weeks, gp100:209-217(210M) + HPV 16 E7:12-20)
Number analyzed (Participants) | 14 | 15
% of CD8+ T cells
  pre-treatment %gp100 g209-2M-specific T cells | 0.02 [0.01 to 0.03] | 0.01 [0.00 to 0.02]
  Post-treatment % gp100 g209-2M-specific T cells | 0.97 [0.37 to 1.57] | 0.98 [0.04 to 1.92]
  Pre-Treatment % HPV16:E7 12-20-specific T cells | 0.61 [0 to 1.27] | 0.1 [0.04 to 0.16]
  Post-Treatment % HPV16:E7 12-20-specific T cells | 0.68 [0.31 to 1.05] | 1.34 [0.85 to 1.82]
Statistical Analysis 1: Comparison: Arm A (Every 2 Weeks, gp100:209-217(210M) and HPV 16 E7:12-20); Test type: Superiority or Other; p < .001, t-test, 2 sided — Post versus Pre-treatment % g209-2M-specific t-cells
Statistical Analysis 2: Comparison: Arm B (Every 3 Weeks, gp100:209-217(210M) + HPV 16 E7:12-20); Test type: Superiority or Other; p < .0001, t-test, 2 sided — Post versus Pre-Treatment %g209-2M-specific T-cells
Statistical Analysis 3: Comparison: Arm A (Every 2 Weeks, gp100:209-217(210M) and HPV 16 E7:12-20) vs Arm B (Every 3 Weeks, gp100:209-217(210M) + HPV 16 E7:12-20); Test type: Superiority or Other; p = 0.59, t-test, 2 sided — Arm A Versus Arm B

ADVERSE EVENTS:
Groups:
- Arm A (Every 2 Weeks): Patients receive gp100:209-217(210M) peptide vaccine and HPV 16 E7:12-20 peptide vaccine mixed with incomplete Freund's adjuvant SC every 2 weeks for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.
  HPV 16 E7:12-20 peptide vaccine: Given SC
  gp100:209-217(210M) peptide vaccine: Given SC
  laboratory biomarker analysis: Correlative studies
- Arm B (Every 3 Weeks): Patients receive gp100:209-217(210M) peptide vaccine and HPV 16 E7:12-20 peptide vaccine mixed with incomplete Freund's adjuvant SC every 3 weeks for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.
  HPV 16 E7:12-20 peptide vaccine: Given SC
  gp100:209-217(210M) peptide vaccine: Given SC
  laboratory biomarker analysis: Correlative studies
Arm/Group | Arm A (Every 2 Weeks) | Arm B (Every 3 Weeks)
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18
Other Adverse Events (participants affected / at risk) | 18/18 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Every 2 Weeks) (N=18) | Arm B (Every 3 Weeks) (N=18)
CVA (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Every 2 Weeks) (N=18) | Arm B (Every 3 Weeks) (N=18)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 18 (18) | 17 (17) — Erythema/Induration/Ecchymosis
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) — Headache/Back/Knee etc
Fatigue (General disorders) | 7 (7) | 13 (13)
Neuropathy (Nervous system disorders) | 3 (3) | 1 (1)
Depression (Nervous system disorders) | 1 (1) | 0 (0)
Endocrine-Other (Endocrine disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Chills (General disorders) | 8 (8) | 6 (6)
Edema (Vascular disorders) | 1 (1) | 2 (2)
Anorexia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dysguesia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (General disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less